CLINICAL TRIAL: NCT00730769
Title: Phase IV.II Pilot Study of Treatment of Cytomegalovirus Infection With a Brief Induction With Ganciclovir i.v. Followed by Valganciclovir Oral in Solid Organ Transplant Patients.
Brief Title: Valganciclovir for Treatment of Cytomegalovirus Infection in Solid Organ Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Salvador Gil-Vernet (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Salvador Gil-Vernet, Nephrologist, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VALGAN-03
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Cytomegalovirus Infection
Keywords: Valganciclovir; Ganciclovir; Pharmacokinetics; Solid organ transplantation; Transplant
MeSH Terms: conditions — Cytomegalovirus Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency | interventions — Ganciclovir; Valganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): Patients received a short induction of IV ganciclovir (Cymevene®; F. Hoffmann-La Roche Ltd, Basel, Switzerland) at 5 mg/kg bid for 5 days (1 hour infusion) , followed by treatment with oral valganciclovir (Valcyte®; F. Hoffmann-La Roche Ltd, Basel, Switzerland) at 900 mg bid (after meals) for 16 days up to complete 21 days of treatment. In patients with impaired renal function, IV ganciclovir and oral valganciclovir doses were adjusted at each visit according to estimated GFR (Cockcroft-Gault equation)
  Interventions: Drug: Single arm (ganciclovir and valganciclovir)

INTERVENTIONS:
Drug: Single arm (ganciclovir and valganciclovir) — Patients received a short induction of IV ganciclovir at 5 mg/kg bid for 5 days (1 hour infusion) , followed by treatment with oral valganciclovir at 900 mg bid (after meals) for 16 days up to complet 21 days of treatment. In patients with impaired renal function, IV ganciclovir and oral valganciclovir doses were adjusted at each visit according to estimated GFR (Cockroft-Gault equation)
  Other Names: Ganciclovir (Cymevene®); Valganciclovir (Valcyte®)

SUMMARY:
The objectives of this study were:

1. To demonstrate the efficacy/safety of a short therapeutic strategy of treatment of CMV infection/disease in SOT patients (kidney, liver and heart recipients) based on 21 days of treatment.
2. To compare the exposure to ganciclovir, at steady state, after oral valganciclovir with respect to ganciclovir given intravenously (i.v.).
3. Evaluate the security of this treatment with valganciclovir.

DETAILED DESCRIPTION:
SOT recipients (kidney, liver and heart transplant) presenting CMV infection or disease were eligible for inclusion if they were ≥18 years of age and presented a positive CMV antigenemia (pp65) defined as ≥ 20positive cells/105 peripherical blood mononuclear cells (PBMC). Patients excluded were those with severe CMV tissue invasive disease, unable to receive oral medication, absolute neutrophil counts less than 500/ mm3, platelets <25000 platelets/mm3, Hemoglobin< 80g/l or estimated glomerular filtration rate< 10 mL/min (according to the Cockcroft-Gault formula).

Patients received a short induction treatment with ganciclovir i.v (Cymevene®; F. Hoffmann-La Roche Ltd, Basel, Switzerland) at the dose of 5 mg/kg/12h, by a peripherical vein infusion of one hour, during 5 days followed by treatment with oral valganciclovir (Valcyte®; F. Hoffmann-La Roche Ltd, Basel, Switzerland) at 900 mg/12h during 16 days, after meals, until complete a total of 21 days of treatment. In patients with impaired renal function ganciclovir i.v. and oral valganciclovir doses were adjusted at each visit according to estimated Glomerular Filtration Rate (GFR) by Cockcroft-Gault equation, as recommended by the manufacturer.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age, solid organ transplant recipients.
* presented a CMV infection demonstrated by CMV antigenemia (pp65) defined as ≥ 20positive cells/105 peripherical blood mononuclear cells (PBMC).
* gave written informed consent.

Exclusion Criteria:

* HIV patients.
* Multiorganic transplant.
* Severe CMV tissue invasive disease.
* Unable to receive oral medication.
* absolute neutrophil counts less than 500/ mm3.
* Platelets <25000 platelets/mm3.
* Hemoglobin< 80g/l.
* Estimated glomerular filtration rate< 10 mL/min (according to the Cockcroft-Gault formula)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-03; Primary Completion 2007-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Dissapeareance of CMV (pp65) antigenemia, determined in peripheral blood mononuclear cells (PBMC). | Baseline, day 5, 10, 15, 21 of treatment and day 30, 60 and 90 of follow-up.

SECONDARY OUTCOMES:
Dissapareance of Cytomegalovirus viremia measured by PCR, determined in plasma samples. | Basal, day 5, 10, 15 and 21 of treatment and 30, 60 and 90 of treatment.
Area under the curve (AUC) of Ganciclovir after ganciclovir i.v. and valganciclovir oral in steady state. | Day 5 (ganciclovir i.v) and day 15 (valganciclovir oral)

CONTACTS AND LOCATIONS:
Overall Officials: Salvador - Gil-Vernet, Medicine, Study Chair — Nephrology Department. Hospital Universitari of Bellvitge
Locations (1):
- Hospital Universitari Bellvitge- Transplant Departments (Liver, Heart and Kidney), L'Hospitalet de Llobregat, Barcelone, Spain

REFERENCES:
- [Derived] Caldes A, Colom H, Armendariz Y, Garrido MJ, Troconiz IF, Gil-Vernet S, Lloberas N, Pou L, Peraire C, Grinyo JM. Population pharmacokinetics of ganciclovir after intravenous ganciclovir and oral valganciclovir administration in solid organ transplant patients infected with cytomegalovirus. Antimicrob Agents Chemother. 2009 Nov;53(11):4816-24. doi: 10.1128/AAC.00085-09. Epub 2009 Sep 8. PMID 19738014